CLINICAL TRIAL: NCT00919724
Title: A Comparison of Endothelial Function Between HIV-infected Subjects Not Receiving Antiretroviral Therapy and Matched HIV-uninfected Control Subjects
Brief Title: Comparing Blood Vessel Endothelial Function in HIV-Infected People and Matched HIV-Uninfected People
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Associate Professor of Medicine, National Heart, Lung, and Blood Institute (NHLBI)
Other Study IDs: 661; R01HL095149 (NIH); HL095149
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infection
Keywords: AIDS; Endothelial Function; Inflammation; Immune Activation; treatment naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HIV-Infected: HIV-infected participants who are not currently receiving antiretroviral medications
- HIV-Uninfected: HIV-uninfected participants matched in age, sex, smoking status, and height to the HIV-infected participants

SUMMARY:
The blood vessels that carry blood from the heart to the rest of the body are normally capable of relaxing and constricting when needed to provide more or less blood to the body. The inability of blood vessels to relax and widen may increase the risk of heart disease and stroke. One potential cause of this inability is inflammation. Because HIV infection is associated with inflammation, it is possible that the blood vessels in people infected with HIV may not relax properly. The purpose of this study is to determine whether people infected with HIV have worse blood vessel function than people without HIV infection.

DETAILED DESCRIPTION:
Normally the insides of blood vessels either widen or narrow in response to the need for more or less blood flow. This is a function of the endothelial cells, which are the cells that line the inner layer of blood vessels. However, in some people endothelial function is impaired, which may put them at an increased risk of heart disease and stroke. It is widely assumed that HIV-infected people not yet receiving antiretroviral medications experience more impaired endothelial function than HIV-uninfected people, possibly because of the link between HIV and inflammation. However, no rigorously controlled study has yet to be performed to verify this presumption. It is important to establish whether HIV infection itself, and not the use of antiretroviral medications, is indeed the cause of impaired endothelial function. This study will compare endothelial function in people with HIV who are not already receiving antiretroviral medications and in people without HIV. Specifically, inflammation, immune activation, endothelial activation, and metabolic measures will be compared.

This study will involve two groups of participants. The first group will consist of people with HIV who are enrolling in two other separate HIV studies (NCT00864916 and NCT00796822), one lasting 8 weeks and the other lasting 48 weeks. The second group will consist of people without HIV who are similar to the first group in terms of age, sex, smoking status, and height. All HIV-infected participants will undergo assessments during the study visits of whichever other HIV study they are enrolled in. All HIV-uninfected participants will attend a main study visit that will include the following: a review of medical records and family medical history; measurements of blood pressure, heart rate, weight, temperature, and waist and hip circumferences; blood and urine collection; and a procedure called brachial artery reactivity testing, which is a noninvasive way to measure endothelial function. Some of the HIV-uninfected participants will continue in the study so that any changes in their endothelial function can be assessed. They will attend either two additional study visits at Weeks 4 and 8, which will correspond with one of the HIV studies, or three additional study visits at Weeks 8, 24, and 48, which will correspond with the other HIV study. The additional visits will include repeat testing except for blood and urine collection.

ELIGIBILITY:
Inclusion Criteria for HIV-Infected Group:

* Positive HIV enzyme-linked immunosorbent assay (ELISA) test with confirmatory Western Blot
* Not currently receiving antiretroviral therapy

Inclusion Criteria for HIV-Uninfected Group:

* Negative HIV ELISA test at screening
* Within 10 years of age of the matched HIV-infected participant
* Same sex and current smoking status as the matched HIV-infected participant
* Height within 4 inches of the matched HIV-infected participant

Exclusion Criteria for All Participants:

* Inability to complete written informed consent
* Incarceration at the time of screening or main study visit
* Diagnosed vascular disease (e.g., history of angina pectoris, coronary disease, peripheral vascular disease, cerebrovascular disease, aortic aneurysm, or otherwise known atherosclerotic disease)
* Diagnosed disease or process associated with increased systemic inflammation (e.g., systemic lupus erythematosis, inflammatory bowel diseases, or other collagen vascular diseases); Note: Hepatitis B or C co-infections are not exclusionary
* History of bleeding diathesis, gastrointestinal ulceration or bleeding, cerebrovascular aneurysm or bleeding, or retinal hemorrhage
* Known or suspected cancer requiring systemic treatment within 6 months of screening
* History of diabetes mellitus, as defined by the American Diabetes Association; Note: History of gestational diabetes is not exclusionary
* History of migraine headaches
* History of Raynaud's phenomenon
* History of cardiac arrhythmias or cardiomyopathy
* History of hypothyroidism or hyperthyroidism, even if treated; Note: Use of caffeinated products, except on the mornings of the study visits, is not exclusionary
* Known allergy or intolerance to nitroglycerin
* History of carotid bruits
* Creatinine clearance less than 50mL/min, using a serum creatinine level measured at screening
* Hemoglobin level greater than 9.0g/dL at screening
* Alanine aminotransferase (ALT) level or aspartate aminotransferase (AST) greater than three times the upper limit of normal (ULN) at screening
* Total bilirubin greater than 2.5 times ULN at screening
* Fever, defined as a temperature greater than 38.0 C within 48 hours prior to screening
* Received therapy for acute infection or other serious medical illness within 14 days prior to screening
* Pregnant or breastfeeding during the course of the study
* Hypotension, defined as systolic blood pressure less than 90mm Hg, at screening.
* Uncontrolled hypertension
* Receipt of anti-inflammatory agents (e.g., plaquenil, infliximab, etanercept, mycophenolate mofetil, sirolimus, tacrolimus, cyclosporine, pentoxifylline, thalidomide)
* Receipt of investigational agents, cytotoxic chemotherapy, systemic or topical glucocorticoids (of any dose), or anabolic steroids within 28 days of screening; Note: Physiologic testosterone replacement therapy is not exclusionary
* Receipt of lipid-lowering drugs, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs), acetazolamide, anticoagulants, anticonvulsants, or thyroid replacements within 7 days prior to screening
* Use of sildenafil, vardenafil, or tadalafil within 72 hours (before or after) of each main study visit
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected people will be recruited from infectious diseases outpatient clinics of Wishard Hospital and Indiana University Hospital. They will be enrolled in one of two other HIV trials. HIV-uninfected people will be recruited from the Indianapolis general population.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K. Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Infectious Diseases Research Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV-Infected | HIV-Uninfected
Started | 45 | 44
Completed | 45 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-Infected | HIV-Uninfected | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [27 to 44] | 35 [25 to 45] | 35 [26 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 35 | 33 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 14 | 42
  White | 17 | 30 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function (Brachial Artery Reactivity)
Description: The maximum change in brachial artery diameter after induction of reactive hyperemia post-release of vascular occlusion. This is a measure of the ability of the endothelium to respond appropriately to lack of tissue oxygenation distal to the point of brachial artery compression.
Time Frame: Single measurement
Measure: Mean (Standard Deviation); unit: percent dilation
Arm/Group | HIV-Infected | HIV-Uninfected
Number analyzed (Participants) | 45 | 44
percent dilation | 3.98 (2.95) [1.91 to 4.99] | 3.37 (2.74) [1.20 to 4.59]
Statistical Analysis 1: Comparison: HIV-Infected vs HIV-Uninfected; Test type: Superiority or Other; p = 0.10, Regression, Linear — Comparison between HIV-infected and HIV-uninfected groups. Comparison adjusted for age, gender, race, height, and brachial artery baseline diameter; Mean Difference (Final Values) = 0.99, Standard Error of Mean 0.60

ADVERSE EVENTS:
Arm/Group | HIV-Infected | HIV-Uninfected
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No